CLINICAL TRIAL: NCT00838630
Title: A Randomized, Two-Way, Single-Dose, Open-Label Study to Evaluate the Bioequivalence of a Test Tablet Formulation of Cilostazol, 100 mg, Compared to an Equivalent Dose of a Commercially Available Reference Drug Product in 36 Fasted, Healthy, Adult Subjects
Brief Title: Cilostazol 100 mg Tablet Formulations Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 03261
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Results first posted 2009-07-21 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Cilostazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Cilostazol 100 mg tablets
- 2 (Active Comparator)
  Interventions: Drug: Pletal® 100 mg tablets

INTERVENTIONS:
Drug: Cilostazol 100 mg tablets — 1 x 100 mg
  Arms: 1
Drug: Pletal® 100 mg tablets — 1 x 100 mg
  Arms: 2

SUMMARY:
The objective of this randomized, single-dose, two-way evaluation is to compare the bioequivalence of a test cilostazol formulation to an equivalent oral dose of the commercially available cilostazol in a test population of 36 adult subjects under fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Sex: Male and Female; similar proportion of each preferred. Female subjects must be surgically sterile for at least six (6) months or postmenopausal for at least one (1) year.
* Age: At least 18 years.
* Weight: Body Mass Index (BMI) of 30 or less.
* Qualifying subjects must be in good health and physical condition as determined by medical history, complete physical examination, and laboratory test, all obtained within four (4) weeks prior to study start. The subject may not have a history of significant past illness expected to affect the investigation. The normal status of subjects will be confirmed by the following procedures:
* Laboratory Tests:

Hemoglobin, hematocrit, RBC, WBC, differential count, serum electrolytes (Na, K, Cl), fasting blood glucose, BUN, bilirubin, creatinine, AST, ALT, LD, alkaline phosphatase, and urinalysis. HIV, Hepatitis B, Hepatitis C, and drugs of abuse testing will be done for screening purposes only. Urine drugs of abuse testing will be repeated at each check-in. Female subjects will have a serum pregnancy test done at screening and a urine pregnancy test prior to each study period at check-in.

Laboratory values which are greater than 20% of the normal range will not qualify unless specifically accepted (with comment) by the Principal Investigator. Results of HIV, Hepatitis B, Hepatitis C, and drugs of abuse must be negative or non-reactive for the subject to qualify for the study.

* Electrocardiogram A 12-lead electrocardiogram (ECG) will be obtained for all subjects. The original tracings, plus interpretation, will be included in the case report form packet.
* Subjects must read and sign the Consent Form.

Exclusion Criteria:

* History of treatment for alcoholism, substance abuse, or drug abuse within past 24 months.
* History of sensitivity to cilostazol, quinolones, or any antiplatelet drug.
* History of malignancy, stroke, diabetes, cardiac, renal or liver disease or other serious illness.
* History of GERD (gastroesophageal reflux disease), malabsorption syndrome, colon cancer, or chronic colitis, including Crohn's disease.
* History of treatment for pulmonary obstruction or asthma within the past five (5) years.
* History of severe headaches or migraines.
* History of glaucoma.
* History of chronic infectious disease.
* History of psychiatric disorder.
* History of thyroid disorder/disease.
* History of hypertension.
* Females who are capable of becoming pregnant or are lactating.
* Inability to read and/or sign the consent form.
* Treatment with any other investigational drug during the four (4) weeks prior to the initial dosing for this study.
* Subjects who have donated blood within four (4) weeks prior to the initial dosing for this study.
* Subjects who smoke or use tobacco products or are currently using nicotine products (patches, gums, etc.). Three months abstinence is required.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2003-11; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Herrmann, M.D., Ph. D., Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Gateway Medical Research Inc., Saint Charles, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cilostazol (Test) First: Cilostazol 100 mg Tablets (test) dosed in first period followed by Pletal® 100 mg Tablets (reference) dosed in second period.
- Pletal® (Reference) First: Pletal® 100 mg Tablets (reference) dosed in first period followed by Cilostazol 100 mg Tablets (test) dosed in second period
Period: First Intervention
Arm/Group | Cilostazol (Test) First | Pletal® (Reference) First
Started | 18 | 18
Completed | 17 | 18
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Washout: 7 Days
Arm/Group | Cilostazol (Test) First | Pletal® (Reference) First
Started | 17 | 18
Completed | 16 | 18
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: Second Intervention
Arm/Group | Cilostazol (Test) First | Pletal® (Reference) First
Started | 16 | 18
Completed | 16 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cilostazol (Test) First | Pletal® (Reference) First | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 16 | 15 | 31
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 17 | 15 | 32
  Black | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 96 hour period
Population: Data from subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cilostazol: Cilostazol 100 mg Tablets (test) dosed in either period
- Pletal®: Pletal® 100 mg Tablets (reference) dosed in either period
Arm/Group | Cilostazol | Pletal®
Number analyzed (Participants) | 34 | 34
ng/mL | 536 (147) | 543 (145)
Statistical Analysis 1: Comparison: Cilostazol vs Pletal®; Test type: Non-Inferiority or Equivalence — Analysis of Variance (ANOVA) will be performed for the log-transformed AUC0-t, AUC0-inf and Cmax parameters; Geometric Test/Ref Ratio x 100 = 98.27, 90% CI [92.32 to 104.61] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 96 hour period
Population: Data from subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cilostazol | Pletal®
Number analyzed (Participants) | 34 | 34
ng*h/mL | 8670 (3626) | 8974 (3147)
Statistical Analysis 1: Comparison: Cilostazol vs Pletal®; Test type: Non-Inferiority or Equivalence — Analysis of Variance (ANOVA) will be performed for log-transformed AUC0-t, AUC0-inf, and Cmax parameters; Geometric Test/Ref Ratio x 100 = 94.37, 90% CI [90.47 to 98.43] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 96 hour period
Population: Data from subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cilostazol | Pletal®
Number analyzed (Participants) | 34 | 34
ng*h/mL | 8430 (3507) | 8634 (3104)
Statistical Analysis 1: Comparison: Cilostazol vs Pletal®; Test type: Non-Inferiority or Equivalence — Analysis of Variance (ANOVA) will be performed on log-transformed AUC0-t, AUC0-inf and Cmax parameters; Geometric Test/Ref Ratio x 100 = 95.70, 90% CI [91.52 to 100.08] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.